CLINICAL TRIAL: NCT01766362
Title: Incidence of Macular Edema After Panretinal Photocoagulation (PRPC) Performed in a Single Session Versus Four Sessions in Diabetic Patients.
Acronym: Pascal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Creuzot Innov 2010
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Type 1 or 2 With Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A session (Experimental)
  Interventions: Procedure: PRPC using Pascal laser
- Four sessions (Other): Every session are spaced out of month
  Interventions: Procedure: PRPC using Pascal laser

INTERVENTIONS:
Procedure: PRPC using Pascal laser

SUMMARY:
The aim of this study is to show that PRPC performed in a single session using a Pascal laser leads to better management of the disease (better rate of regression of neovessels, lower risk of a loss of visual acuity in the long term related to macular edema), a saving of time and better comfort for both patient and doctor.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 1 or 2
* Subjects with severe non-proliferative or early proliferative diabetic retinopathy (according to the Alfediam classification)
* Subjects with central macular thickness less than or equal to 350 µm according to spetralis OCT
* Subjects registered with a social security agency
* Subjects who have provided written informed consent
* Subjects aged 18 or above

Exclusion Criteria:

* Pregnancy
* Breastfeeding women
* Patients presenting a contra-indication to Mydriaticum and Neosynephrine
* History of glaucoma or non-controlled ocular hypertension
* Blindness in one eye
* History of renal insufficiency requiring dialysis, or kidney or pancreas transplantation
* Unbalanced diabetes requiring, in the previous 4 months, intensive insulin therapy.
* Central macular thickness greater than 350 µm
* Visual acuity less than 20/32 measured using an ETDRS chart
* Proliferative diabetic retinopathy associated with "high risk factors" (extensive prepapillary neovessels and/or preretinal or prepapillary neovessels associated with preretinal of intravitreal hemorrhage)
* Macular edema due to causes other than diabetic retinopathy (venous occlusion, uveitis) or occurring in a context of vitreomacular traction
* Already started PRPC
* History of eye surgery or YAG laser capsulotomy performed during the preceding 6 months
* Subjects under legal supervision or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Macular thickness | 9 months after the start of traitement
  Central macular thickness at 9 months after the start of PRPC using Pascal laser.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU Dijon, Dijon
  - CHU de la Croix Rousse, Lyon
  - Hôpital Lariboisière, Paris

REFERENCES:
- [Result] Gabrielle PH, Massin P, Kodjikian L, Erginay A, Pallot C, Jonval L, Soudry A, Couturier A, Vardanian-Vartin C, Bron AM, Creuzot-Garcher C. Central retinal thickness following panretinal photocoagulation using a multispot semi-automated pattern-scanning laser to treat ischaemic diabetic retinopathy: Treatment in one session compared with four monthly sessions. Acta Ophthalmol. 2019 Aug;97(5):e680-e687. doi: 10.1111/aos.14002. Epub 2018 Dec 18. PMID 30561087